CLINICAL TRIAL: NCT00356473
Title: Effects of Atorvastatin on Disease Activity and HDL Cholesterol Anti-inflammatory Properties in Patients With Rheumatoid Arthritis
Brief Title: Effects of Atorvastatin on Disease Activity and HDL Cholesterol Function in Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 02-07-061-02
Record Dates: First submitted 2006-07-25; First posted 2006-07-26 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2006-06

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; Atherosclerosis; High density lipoprotein (HDL) cholesterol; Statins; HDL anti-inflammatory properties; Atorvastatin
MeSH Terms: conditions — Arthritis, Rheumatoid; Atherosclerosis | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Atorvastatin
- Atorvastatin (Experimental): Atorvastatin
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin

SUMMARY:
This research evaluates the effects of a cholesterol-lowering medication, atorvastatin, on both arthritis activity and the ability of high-density lipoprotein cholesterol (HDL-C, sometimes referred to as "good cholesterol") to prevent changes in low-density lipoprotein cholesterol (LDL-C, sometimes referred to as "bad cholesterol"), which lead to atherosclerosis, or "hardening of the arteries." We hypothesize that atorvastatin may improve both joint inflammation and the anti-inflammatory properties of HDL cholesterol.

DETAILED DESCRIPTION:
Heart attacks are the leading cause of death in patients with rheumatoid arthritis (RA). Cardiovascular events occur more frequently than would be expected in patients with RA and traditional heart risk factors do not explain this increased risk. Further research is needed to pursue ways of reducing heart disease mortality and improving outcome in patients with RA.

There is reason to believe that a class of cholesterol-lowering medications called statins, beneficial in cardiovascular disease prevention, may be able to reduce the irritation of the joints ("inflammation") associated with RA. Statins have been shown to reduce manifestations of inflammation in the blood of patients at increased risk for heart disease, and in the process reduce the risk of heart attack, stroke, and sudden death. Some similarities in the nature of both RA and heart disease may suggest potential benefits of statin therapy in both conditions.

In addition to inflammation, another factor which may contribute to coronary heart disease (CHD) risk in RA patients is dysfunctional high-density lipoprotein cholesterol (HDL-C, sometimes referred to as "good cholesterol"). Normally, HDL-C acts to counter a type of damage called "oxidation" within LDL-C which is a critical step in the development and progression of heart disease. Data from patients with RA and system lupus erythematosus (SLE) suggests that patients with active rheumatic diseases such as RA and SLE may have increased amounts of dysfunctional HDL-C, and therefore they may be at increased risk of heart disease. A blood test developed by Dr. Navab and colleagues at UCLA rapidly assesses this HDL-C function. This study will investigate both the level of HDL-C antioxidant function in patients with active RA as well as whether abnormal HDL function can be improved by statin use in this population. This research also evaluates the effects of atorvastatin on arthritis activity. We hypothesize that atorvastatin may improve both joint inflammation and the anti-inflammatory properties of HDL cholesterol.

ELIGIBILITY:
Inclusion Criteria:

Fulfill American College of Rheumatology (ACR) criteria for RA

At least 18 years of age

Have RA for at least one year with ongoing active disease (active disease defined as at least two of three: 1) ≥ six tender joints; 2) ≥ three swollen joints; 3) ≥ 45 minutes of morning stiffness)

Taking stable doses of disease modifying anti-rheumatic drug (DMARD) therapy for at least 3 months prior to study entry -

Exclusion Criteria:

Unable to give informed consent

Pregnant or lactating

Eligible for pharmacologic lipid-lowering therapy per National Cholesterol Treatment Program Adult Treatment Panel III guidelines

Using any lipid lowering medication

Known hepatic disease

Elevated liver transaminase levels within the past two months

Previous treatment in the last three months with hydroxychloroquine

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2003-03; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
HDL anti-inflammatory properties at 0 and 12 weeks | at 0 and 12 weeks
Highly sensitive C-reactive protein (hs-CRP) at 0 and 12 weeks | at 0 and 12 weeks

SECONDARY OUTCOMES:
Disease activity score using a 28 joint count (DAS28) at 0,3,6,12, and 18 weeks | at 0,3,6,12, and 18 weeks
Patient and physician global assessments on visual analogue pain scale (VAS; 0-100) at 0,3,6,12, and 18 weeks | at 0,3,6,12, and 18 weeks
Swollen and tender joint counts at 0,3,6,12,and 18 weeks | at 0,3,6,12, and 18 weeks
Patient pain assessment on VAS (0-100)at 0,3,6,12, and 18 weeks | at 0,3,6,12, and 18 weeks
Erythrocyte sedimentation rate(Westergren) at 0,3,6,12, and 18 weeks | at 0,3,6,12, and 18 weeks
Cholesterol levels at 0,3,6,12, and 18 weeks | at 0,3,6,12, and 18 weeks
Health assessment questionnaire disability index (HAQ-DI) at 0,3,6,12, and 18 weeks | at 0,3,6,12, and 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin J Ansell, MD, Principal Investigator — University of California, Los Angeles

REFERENCES:
- [Derived] Charles-Schoeman C, Khanna D, Furst DE, McMahon M, Reddy ST, Fogelman AM, Paulus HE, Park GS, Gong T, Ansell BJ. Effects of high-dose atorvastatin on antiinflammatory properties of high density lipoprotein in patients with rheumatoid arthritis: a pilot study. J Rheumatol. 2007 Jul;34(7):1459-64. Epub 2007 Jun 1. PMID 17552046